CLINICAL TRIAL: NCT00689299
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Ranging Study of Sublingual Immunotherapy (SLIT) in Adults Sensitized to the Standardized Allergenic Extract, Cat Hair (Felis Domesticus)
Brief Title: Phase 2 Study in Adults Sensitized to Cat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antigen Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALI002-08; ALI002-08 (Other: Antigen Laboratories, Inc.)
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Allergy
Keywords: Sublingual Immunotherapy (SLIT); Non-seasonal allergic rhinitis; Immunotherapy; Allergic rhinitis; Cat; Perennial allergy; Non-seasonal allergy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic, Perennial; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Group C (Placebo Comparator): Standardized Allergenic Extract, Cat Hair (Felis domesticus) placebo
  Interventions: Biological: Placebo
- Dose Group A (Active Comparator): Standardized Allergenic Extract, Cat Hair (Felis domesticus) 0.21 Units
  Interventions: Biological: Standardized Allergenic Extract, Cat Hair
- Dose Group B (Active Comparator): Standardized Allergenic Extract, Cat Hair (Felis domesticus)2.1 units
  Interventions: Biological: Standardized Allergenic Extract, Cat Hair

INTERVENTIONS:
Biological: Standardized Allergenic Extract, Cat Hair — Standardized Cat Hair Allergenic Extract sublingual drops
  Other Names: Standardized Cat Hair Allergenic Extract
  Arms: Dose Group A; Dose Group B
Biological: Placebo — Placebo Sublingual Drops
  Arms: Dose Group C

SUMMARY:
The purpose of this study is to identify an effective dose of allergen-specific immunotherapy for cat hair (Felis domesticus) administered by the oral/sublingual route.

DETAILED DESCRIPTION:
This was a phase 2, randomized, double-blind, placebo-controlled, parallel groups study conducted in 3 centers in the US (NCT00689299). Study drug was sublingually dosed once daily as 0.15 mL of US standardized cat hair extract dosed either undiluted, as 1:10 dilution, or placebo. Target dose was obtained on Day 3 of dose titration escalating through 1:100 and 1:10 dilutions on Day 1 and Day 2 in the high dose group or placebo and 1:100 dilutions in the low dose group. Treatment duration was 20 weeks. Adult (>18 years) study subjects had positive history for cat allergy without asthma, positive skin test to cat allergen, absence of immunotherapy during the prior 2 years, and absence of other confounding baseline conditions. The primary outcome parameter was average Total Symptom Score (TSS) during a 1-hour cat chamber exposure. TSS is the sum of 7 items rated from 0 - 3 (none to severe) for nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) and non-nasal symptoms (eye watering, eye itching, and itching palate/ ear/ throat).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages of 18 and 55 years (inclusive).
* Written informed consent to participate in the study.
* Documented allergy to cat hair as demonstrated by a positive epicutaneous skin test (wheal >3 mm) and symptoms of allergic rhinitis during exposure to cats.
* Female subjects of childbearing potential, defined as not surgically sterile or at least 2 years postmenopausal, must agree to use one of the following forms of contraception from screening through the 4 week follow-up period following the last dose of clinical trial: hormonal begun >30 days prior to screening, barrier, intrauterine device or vasectomized partner (6 months minimum).
* No clinically significant abnormal findings on physical examination, with the exception of head, ears, eyes, nose, and throat (HEENT) findings consistent with allergic rhinitis, medical history, or clinical laboratory results during screening which would jeopardize the safety of the subject or impact validity of study results.

Exclusion Criteria:

* Previous allergen immunotherapy (subcutaneous immunotherapy (SCIT), oral immunotherapy, sublingual immunotherapy (SLIT) or recombinant peptide) for cat within 24 months of Screening Visit.
* History of severe allergic reaction requiring medical intervention.
* Intolerance of or severe allergic reaction to previous immunotherapy (SCIT, oral immunotherapy, SLIT, or recombinant peptide).
* Allergy to any of the non-antigen ingredients in the study drug formulation, including, but not limited to: Food, Drug and Cosmetic Act (FD&C) Yellow #5, Red #40 and Blue #1; sodium chloride; sodium bicarbonate; and glycerine.
* History of asthma requiring daily medication.
* Subjects receiving anti-IgE monoclonal antibodies.
* Congenital immune deficiency or acquired immune suppression. Causes of acquired immune suppression may include, but are not limited to, systemic illnesses such as malignancy and infection, the use of medications such as corticosteroids and chemotherapeutic agents, and radiation therapy.
* History of organ transplant, hematologic malignancy, autoimmune disease, myocardial infarction, or congestive heart failure.
* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, psychiatric, or cardiovascular disease, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Inability or unwillingness to stop using drugs that may inhibit the wheal-and-flare reaction or rhinitic response prior to the study and for the duration of dosing clinical trial material (CTM), with the exception of protocol-specified rescue medications provided by the study site for use after Study Day 0. This includes, but is not limited to:

  * Decongestants for 3 days prior to Study Day 0
  * H1 antagonists (antihistamines) (oral, nasal or ocular) for 7 days prior to Study Day 0
  * Topical intranasal corticosteroids for 14 days prior to Study Day 0
  * Cromolyn or nedocromil for 14 days prior to Study Day 0
  * Systemic corticosteroids for 28 days prior to Study Day 0
  * Tricyclic antidepressants for 28 days prior to Study Day 0
  * Leukotriene modifiers for 7 days prior to study Day 0
* Inability or unwillingness to stop using drugs that may inhibit the ability to treat a severe allergic adverse event. This includes, but is not limited to: beta blockers such as atenolol (Tenormin®), metoprolol (Lopressor®, Toprol-XL®) and propranolol (Inderal®, Inderal LA®) for 14 days prior to Study Day 0 and for the duration of the study.
* Female subjects who are trying to conceive, are pregnant, or are lactating.
* Positive serum pregnancy test at screening or a positive human chorionic gonadotropin (HCG) urine test on Study Day 0 prior to administration of study drug for women of childbearing potential.
* Positive blood screen for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbSAg), or Hepatitis C.
* Forced Expiratory Volume in 1 second (FEV1) <70% of the predicted value.
* History of alcohol or drug abuse within the year prior to the Screening Visit, or current evidence of substance dependence or abuse.
* Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to the Screening Visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Berkowitz, M.D., Principal Investigator — Allergen Response Research Center
Locations (3):
- United States (3):
  - Allergy & Asthma Medical Group & Research Center, San Diego, California
  - Allergen Response and Research Center, Marietta, Georgia
  - Clinical Research Center, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Maintenance dose of 0.15 mL of liquid placebo administered as a daily oral liquid via sublingual route.
- 2.1 Units Fel d 1: Active Dose Group B
  From a concentration of 14.0 Units/mL of Fel d 1, a maintenance dose of 0.15 mL (2.1 Units Fel d 1) was administered as a daily oral liquid via sublingual route.
- 0.21 Units Fel d 1: Active Dose Group A
  From a concentration of 14.0 Units/mL of Fel d 1 diluted 1:10 v/v, a maintenance dose of 0.15 mL (0.21 Units Fel d 1) was administered as a daily oral liquid via sublingual route.
Period: Overall Study
Arm/Group | Placebo | 2.1 Units Fel d 1 | 0.21 Units Fel d 1
Started | 58 | 57 | 54
Completed | 51 | 54 | 49
Not Completed | 7 | 3 | 5
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo - Dose Group C
- 0.21 Units Fel d 1 Standardized Allergenic Extract, Cat Hair (: Active Dose Group A
- 2.1 Units Fel d 1 Standardized Allergenic Extract, Cat Hair (F: Active Dose Group B
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.21 Units Fel d 1 Standardized Allergenic Extract, Cat Hair ( | 2.1 Units Fel d 1 Standardized Allergenic Extract, Cat Hair (F | Total
Number analyzed (Participants) | 58 | 54 | 57 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 58 | 54 | 57 | 169
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9) | 36 (8) | 33 (9) | 34.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 33 | 38 | 110
  Male | 19 | 21 | 19 | 59
Region of Enrollment [Number; unit: participants]
  United States | 58 | 54 | 57 | 169

OUTCOME MEASURES:

1. Primary Outcome: Scores on a Scale (Average of Total Symptom Scores)
Description: Sum of individual symptoms scores, 7 items, 21 points maximum
  Total Symptom Scores during environmental chamber exposures at week 20. The Total Symptom Score was defined as the sum of the scores from the following seven symptoms rated 0-3 (0=absent, 1=mild, 2= moderate, 3=severe): runny nose, sneezing, itching nose, nasal congestion, watery eyes, itchy eyes, and itchy ears/palate/throat.
  Total Symptom score could range from 0-21; the lower the score, the more favorable the outcome. Each symptom parameter was graded by the study subject every 10 minutes for up to 60 minutes during the baseline (Day 0) and during the Week 20 environmental chamber exposures.
Time Frame: 20 weeks
Population: Modified Intent to Treat. All subjects with at least 1 symptom assessment during post treatment chamber exposure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo: Dose Group C: placebo Standardized Allergenic Extract, Cat Hair (Felis domesticus)
- 0.21 Units Standardized Allergenic Extract, Cat Hair: Dose Group A
- 2.1 Units Standardized Allergenic Extract, Cat Hair: Dose Group B
Arm/Group | Placebo | 0.21 Units Standardized Allergenic Extract, Cat Hair | 2.1 Units Standardized Allergenic Extract, Cat Hair
Number analyzed (Participants) | 58 | 54 | 57
Scores on a scale | 7.02 (4.48) | 8.30 (5.14) | 7.87 (4.99)
Statistical Analysis 1: Comparison: Placebo vs 0.21 Units Standardized Allergenic Extract, Cat Hair vs 2.1 Units Standardized Allergenic Extract, Cat Hair; ANOVA with baseline score as covariate; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 20 weeks treatment plus 30 days post treatment followup.
Description: Both SAEs reported in this study occurred in the 30 day post treatment followup, and were classified as not treatment related.
Groups:
- Dose Group C: placebo Standardized Allergenic Extract, Cat Hair (Felis domesticus)
- Dose Group A: 0.21 Units Standardized Allergenic Extract, Cat Hair (Felis domesticus)
- Dose Group B: 2.1 Units Standardized Allergenic Extract, Cat Hair (Felis domesticus)
Arm/Group | Dose Group C | Dose Group A | Dose Group B
Serious Adverse Events (participants affected / at risk) | 0/58 | 2/54 | 0/57
Other Adverse Events (participants affected / at risk) | 26/58 | 20/54 | 33/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group C (N=58) | Dose Group A (N=54) | Dose Group B (N=57)
Severe headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group C (N=58) | Dose Group A (N=54) | Dose Group B (N=57)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 16
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Lacrimation increased (Eye disorders) | 3 | 4 | 2
Eye pruritus (Eye disorders) | 3 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8 | 11
Nausea (Gastrointestinal disorders) | 4 | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4
Oral pruritus (Gastrointestinal disorders) | 2 | 1 | 5
Paraesthesia oral (Gastrointestinal disorders) | 3 | 2 | 2
Ear pruritus (Ear and labyrinth disorders) | 2 | 4 | 8

LIMITATIONS AND CAVEATS:
Adverse events: 41%, 58%, and 45% > 5% in Group A, B, and C, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No